CLINICAL TRIAL: NCT06219499
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Immunogenicity and Pharmacokinetics of ONC-841 When Administered Intravenously in Healthy Adult Subjects
Brief Title: Safety, Tolerability, Immunogenicity and Pharmacokinetics of ONC-841
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA reviewers asked for Phase 1 study in Oncology subjects, not in healthy volunteers.
Sponsor: OncoC4, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ONC-841-001
Record Dates: First submitted 2023-12-29; First posted 2024-01-23 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- ONC-841 (Experimental)
  Interventions: Drug: ONC-841

INTERVENTIONS:
Drug: ONC-841 — ONC-841 is a humanized monoclonal antibody.
  Arms: ONC-841
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The Phase 1 study is a randomized, double-blind, placebo-controlled, single ascending dose, multi-cohort study. The study will evaluate 5 dose levels of the investigational product, in 5 cohorts of 8 healthy volunteers per cohort. In each cohort, 6 volunteers will receive the investigational product and 2 volunteers will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adult males and females, 18 to 55 years of age (inclusive) at screening.
3. Body mass index ≥ 18.0 and ≤ 30.0 kg/m2, with a body weight (to 1 decimal place) ≥ 50 kg at screening.
4. Be non-smokers (including tobacco, e-cigarettes and marijuana) for at least 3 months prior to first study drug administration and have a negative test for cotinine at the screening visit and at check- in on Day -1.
5. Medically healthy without clinically significant abnormalities (in the opinion of the PI) at the screening visit and prior to dosing at the timepoints indicated in the Schedules of Assessments (SoA), including:

   1. Physical examination without any clinically significant findings;
   2. Systolic blood pressure in the range of 90 to 140 mmHg (inclusive) and diastolic blood pressure in the range of 40 to 90 mmHg (inclusive) after 5 minutes in supine (or semi- supine) position;
   3. Heart rate in the range of 40 to 100 bpm (inclusive) after 5 minutes rest in supine (or semi- supine) position;
   4. Body temperature (tympanic or oral) in the range 35.5°C to 37.5°C (inclusive);
   5. No clinically significant findings in serum chemistry, haematology, coagulation, and urinalysis tests (any of the routine laboratory test may be repeated at the discretion of the PI);
   6. Triplicate 12-lead ECG (taken after the volunteer has been supine (or semi-supine) for at least 5 minutes) with a QT interval corrected using the Fridericia method (QTcF) ≤ 450 msec for males and ≤ 470 msec for females and no clinically significant abnormalities.
6. Female volunteers must:

   a. Be of nonchildbearing potential i.e., be surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before screening) or be postmenopausal, where menopause is defined as 12 months of amenorrhea in the absence of other biological causes. Females under the age of 55 years must have a documented serum follicle-stimulating hormone (FSH) level > 40mIU/mL to confirm menopause (females who are taking Hormone Replacement Therapy (HRT) should provide evidence that they are post-menopausal or should be excluded as their post-menopausal status cannot be confirmed by measuring FSH - alternatively they would need to stop HRT to allow FSH to be measured).

   b. If of childbearing potential (defined as any female who has experienced menarche and who has not undergone surgical sterilisation and is not postmenopausal), the participant:
   * Must have a negative serum test at the screening visit and a negative urine pregnancy test within 24 hours prior to the start of study drug;
   * Must not be breastfeeding, lactating or planning pregnancy during the study period;
   * Must agree not to attempt to become pregnant;
   * If not exclusively in same-sex relationships, must agree to use adequate contraception (which is defined as use of a condom by the male partner combined with use of a highly effective method of contraception by the female partner; refer to Appendix 5. Highly Effective Forms of Contraception) after signing consent, during the study, and at least 30 days after the EoS visit;
   * Must agree to not donate ova for at least 30 days after the EoS visit.
7. Male participants, if not surgically sterilised, must agree to:

   1. Not donate sperm after signing consent, during the study, and at least 90 days after the EoS visit;

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the past 3 months determined by the PI to be clinically significant (participants with resolved childhood asthma may be included in the study).
2. Current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic or antiviral medications.
3. Suffer from frequent or recurrent infections (defined as ≥3 occurrences in the 12 months preceding first study drug administration or 2 occurrences in the 6 months preceding first study drug administration).
4. Any history of malignant disease in the last 10 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
5. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia.
6. Use of or plans to use systemic immunosuppressive (e.g., corticosteroids, methotrexate, azathioprine, cyclosporine) or immunomodulating medications (e.g., interferon) during the study or within 3 months prior to the first study drug administration (prior use of nasal sprays for hayfever may be permitted if used > 30 days prior to study drug administration or alternatively at the discretion of the PI).
7. History of risk factors for torsade de pointes (including a family history of long QT syndrome or sudden cardiac death) or a known arrythmia.
8. Liver function test results elevated more than 1.5-fold above the upper limit of normal (ULN) for gamma glutamyl transferase (GGT), bilirubin (total, conjugated and unconjugated), alkaline phosphatase (ALP), aspartate aminotransferase (AST) or alanine aminotransferase (ALT). Volunteers with ALP and/or ALT/AST above the limits specified may be included, at the discretion of the PI, if the levels are unaccompanied by clinical signs and are determined to be normal variants.
9. Positive test results for active human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or Quantiferon Gold® (Tuberculosis (TB) infection) at the screening visit.
10. Presence or having sequelae of gastrointestinal, liver, kidney, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs (prior gall bladder and/or appendix removal is not exclusionary if the procedure was undertaken ≥ 3 months prior to study drug administration; if less than 3 months, history of such procedures may still be considered not exclusionary if it is deemed appropriate by the PI).
11. Estimated creatinine clearance (CrCl) < 60 mL/min using the Cockcroft-Gault formula or serum creatinine more than 1.5-fold above the ULN.

History of substance abuse or alcohol abuse within 12 weeks prior to the screening visit (defined as more than an average of 14 standard drinks per week or regular consumption of more than 4 standard drinks on any one day; where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc./Vol], 100 mL wine [12% Alc./Vol], 30 mL spirit [40% Alc./Vol]).

13. Positive drugs of abuse or alcohol breath test results at the screening visit or at check-in (Day -1).

14. Use of any prescription or over-the-counter medication (including herbal products, and hormone supplements) within 10 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration - exceptions include occasional use of paracetamol (doses of 500 mg up to every 6 hours or 2 g per day maximum for no more than 3 consecutive days), ibuprofen (doses of 400 mg up to every 6 hours or 1.2 g per day maximum for no more than 3 consecutive days), topical ointments, and vitamins or dietary supplements.

15. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the PI, would interfere with the volunteer's ability to participate in the trial.

16. Known hypersensitivity to any of the study drug ingredients. 17. Use of any vaccinations within 14 days (within 4 weeks for live virus vaccines) prior to the first study drug administration.

18. For women of childbearing potential, a positive serum pregnancy test at the screening visit or a positive urine pregnancy test (with confirmatory serum pregnancy test) at check-in (Day -1).

19. Females who are breastfeeding or planning to breast feed at any time during the study.

20. Donation of blood or plasma within 30 days prior to first study drug administration, or loss of whole blood of more than 500 mL within 30 days prior to first study drug administration, or receipt of a blood transfusion within 1 year of first study drug administration.

21. Treatment with an investigational drug in another clinical trial within 60 days or 5 half-lives of the other investigational drug (whichever is longer) prior to the first administration of study drug in this trial.

22. Any other condition or prior therapy that in the opinion of the PI would make the volunteer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 42 Days
  The number of subjects who have Dose limiting toxicity (DLT) as defined by protocol DLT criteria during the first cycle of study drug, ONC-841, administration.
Maximum Toxicity Dose (MTD) | 42 Days
  Maximal tolerable dose (MTD), the study drug, ONC-841, dose level that has two out of six subjects who have DLT.

SECONDARY OUTCOMES:
Cmax of ONC-841 | PK samplings in cycle1, pre-dose and post-dose samples, and End of Treatment
  The highest Serum concentration of ONC-841 after IV infusion at cycle 1 and cycle 3 dosings from different timepoints after drug administration.intravenous dose in healthy adult volunteers
The serum half-life of ONC-841 | PK samplings in cycle1, pre-dose and post-dose samples, and End of Treatment
  To determine the drug concentration in serum samples that are taken in various timepoints during the treatment in order to calculate drug half life.